CLINICAL TRIAL: NCT01876966
Title: A Phase I, Partially Randomized, Open Label, Two-way, Two Period Cross-over Study to Investigate the Pharmacokinetic Interaction Between Etravirine or Darunavir/Rtv and Artemether/Lumefantrine at Steady-state in Healthy HIV-negative Subjects
Brief Title: Interaction Between Etravirine or Darunavir/Ritonavir and Artemether / Lumefantrine
Acronym: DDI Coartem
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CR018409; 2010-023289-31 (EudraCT Number); TMC125VIR1001 (Other: Janssen CTMS ID)
Record Dates: First submitted 2012-11-19; First posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: HIV
Keywords: HIV; pharmacokinetic interaction; healthy HIV-negative person
MeSH Terms: interventions — etravirine; Darunavir; Ritonavir; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETR, artemether/lumefantrine (Experimental): treatment with artemether/lumefantrine 80/480 mg during 3 days (treatment A) and treatment during 22 days with etravirine for 22 days and artemether/lumefantrine 80/480 mg from day 8 to day 11 (treatment B) with a washout of at least 4 weeks between the 2 treatment periods
  Interventions: Drug: Etravirine; Drug: artemether/lumefantrine
- DRV/rtv, artemether/lumefantrine (Experimental): treatment with artemether/lumefantrine 80/480 mg during 3 days (treatment A) and treatment during 22 days with darunavir/ritonavir and artemether/lumefantrine 80/480 mg from day 8 to day 11 (treatment B) with a washout of at least 4 weeks between the 2 treatment periods
  Interventions: Drug: Darunavir/ritonavir; Drug: artemether/lumefantrine

INTERVENTIONS:
Drug: Etravirine — 200 mg ETR b.i.d. from Day 1 to Day 21 with a single 200 mg dose of ETR in the morning on Day 22
  Arms: ETR, artemether/lumefantrine
Drug: Darunavir/ritonavir — DRV/rtv 600/100 mg b.i.d. from Day 1 to Day 21 with a single dose of DRV/rtv in the morning on Day 22
  Arms: DRV/rtv, artemether/lumefantrine
Drug: artemether/lumefantrine — 3 days of treatment with artemether/lumefantrine 80/480 mg (6 doses of 4 tablets [20/120 mg] at 0, 8, 24, 36, 48, and 60 hours)

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic interaction between etravirine and artemether/lumefantrine and darunavir/ritonavir and artemether/lumefantrine in healthy Human Immunodeficiency Virus- (HIV-)negative patients. 'Pharmacokinetic interaction' means that one medication can influence the absorption and elimination from the body of the other medication.

DETAILED DESCRIPTION:
This is a Phase I, partially randomized, open-label, single-center, two-way, two-period cross-over study to investigate the pharmacokinetic interaction between etravirine (ETR) or darunavir/ritonavir (DRV/rtv) and the antimalarial drugs artemether/lumefantrine at steady-state in healthy human immunodeficiency virus (HIV)-negative patients. The study population will consist of 32 healthy patients, equally divided over 2 panels. Patients in Panel 1 will be treated with ETR and artemether/lumefantrine; patients in Panel 2 will be treated with DRV/rtv and artemether/lumefantrine. Treatment A will consist of 3 days of treatment with artemether/lumefantrine. Treatment B will consist of 200 mg ETR twice daily (b.i.d.) (Panel 1) or 600/100 mg DRV/rtv b.i.d. (Panel 2) from Day 1 to Day 21 with a single dose of ETR (Panel 1) or DRV/rtv (Panel 2) in the morning on Day 22. From Day 8, 3 days of treatment with artemether/lumefantrine. In a first stage of treatment in Panel 2, only 4 patients will be allowed to start Treatment B. Based on the ECG results of the first 4 patients with evaluable ECG data after assessments on Day 11 (66 hours after the combined intake of DRV/rtv and artemether/lumefantrine), the Sponsor will decide whether additional patients can be allowed to start Treatment B. There will be a washout period of at least 4 weeks between Treatments A and B. Half of the patients of Panel 1 (8 patients) and Panel 2 (8 patients) will be randomized to sequence AB and half will be randomized to sequence BA. Randomization in Panel 2 will occur in two steps. In Step 1, 4 patients will be allocated to sequence BA and evaluated for QTc prolongation. Based on the outcome of their ECG results, the Sponsor will decide whether the remainder of patients will be randomized in Step 2, i.e. 4 patients to BA and 8 patients to AB (1:2 randomization). Serial pharmacokinetic assessments will be determined for Panels 1 and 2 in Treatments A and B for artemether and its metabolite dihydroartemisinin (DHA) after the first intake of artemether/lumefantrine over 8 hours and after the last intake of artemether/lumefantrine over 72 hours (3 days), and for lumefantrine after the last intake of artemether/lumefantrine over 264 hours (11 days). Serial pharmacokinetic assessments will be determined for ETR (Panel 1) or DRV and rtv (Panel 2) over the 12-hour dosing interval on Day 8 (after the morning intake) and Day 11 (after the last dose of artemether/lumefantrine) of Treatment B. All ETR, DRV/rtv and artemether/lumefantrine treatments will be administered under fed conditions and will be taken within 10 minutes after completion of a meal. Safety and tolerability evaluations will be recorded on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

* if of childbearing potential or if male, use a highly effective method of birth control.
* Able to comply with protocol requirements.
* A BMI (weight in kg divided by the square of height in meters) of 18.5 to 30.0 kg/m2, extremes included.
* healthy on the basis of a medical evaluation
* Non-smoking for at least 3 months prior to selection.

Exclusion Criteria:

* previously demonstrated clinically significant allergy, hypersensitivity or intolerance to any of the investigational medications or its excipients
* Use of concomitant medication, including over-the-counter products and dietary supplements.
* Having participated in more than 1 study (single or multiple dose) with ETR (TMC125), DRV (TMC114), dapivirine (TMC120) and/or rilpivirine (TMC278, formerly known as R278474), or having developed a rash, erythema or urticaria while participating in a study with the aforementioned compounds.
* A positive pregnancy test or breast feeding at screening or on Day 1.
* Any condition that, in the opinion of the investigator, would compromise the study or the well-being of the patient or prevent the patient from meeting or performing study requirements

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
effect of ETR or DRV/rtv on the plasma concentrations of artemether, lumefantrine and dihydroartemisinin | Treatment A: Day 1-2 & Day 4-15; Treatment B: Day 8-9 & Day 11-22
  the effect of ETR or DRV/rtv on the pharmacokinetics of artemether, lumefantrine and the artemether metabolite dihydroartemisinin (DHA) after single and multiple dose(s) in healthy subjects. plasma concentrations: minimum (Cmin) and maximum (Cmax): artemether and DHA (Day 11 of Treatment B versus Day 4 of Treatment A, Days 11-14 of Treatment B versus Days 4-7 of Treatment A ), lumefantrine (Days 11-22 of Treatment B versus Days 4-15 of Treatment A ); Cmax artemether and DHA (Day 8-9 of Treatment B versus Day 1-2 of Treatment A )
effect of ETR or DRV/rtv on the Area under the concentration-time curve (AUC) in plasma for artemether, lumefantrine and dihydroartemisinin | Treatment A: Day 1-2 & Day 4-15; Treatment B: Day 8-9 & 11-22
  effect of ETR or DRV/rtv on the AUC from time of administration (0 hours) to 8 hours after dosing (AUC8h): artemether and DHA (Day 8-9 of Treatment B versus Day 1-2 of Treatment A); AUC from 0 to 12 hours (AUC 12h) artemether and DHA (Day 11 of Treatment B versus Day 4 of Treatment A ); AUC from 0 to 264 hours (AUC264h) lumefantrine (Days 11-22 of Treatment B versus Days 4-15 of Treatment A ; AUC from 0 to the last time point with a measurable concentration post dosing (AUClast) artemether and DHA (Days 11-14 of Treatment B versus Days 4-7 of Treatment A )
Plasma concentrations of ETR, DRV and rtv | Treatment B: Day 8 & Day 11
  Cmin and Cmax for ETR, DRV and ritonavir (Day 11 of Treatment B versus Day 8 of Treatment B )
Area under the concentration-time curve (AUC) in plasma for ETR, DRV and rtv | Treatment B: Day 8 & Day 11
  AUC from time of administration to 12 hours after dosing (AUC12h) for ETR, DRV and ritonavir (Day 11 of Treatment B versus Day 8 of Treatment B)

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | at screening, during treatment and at day 7 and 30, 31 or 32 after last study medication intake
  short-term safety and tolerability of coadministration of ETR or DRV/rtv and artemether/lumefantrine in healthy subjects.
Profile of pharmacokinetics of ETR by cytochrome P450 (CYP)2C9 and CYP2C19 genotype | Treatment B: Day 8
  the effect of CYP2C9 and CYP2C19 genotypes will be evaluated by comparison of these genotypes with the Cmax and AUC12 for ETR
Profile of pharmacokinetics of artemether and DHA after single and multiple dose(s) | Treatment A: Day 1-2 & Day 4-7
  Cmax (both periods), AUC8h (Day 1-2) and AUClast (Day 4-7) for artemether and DHA

REFERENCES:
- [Result] Kakuda TN, DeMasi R, van Delft Y, Mohammed P. Pharmacokinetic interaction between etravirine or darunavir/ritonavir and artemether/lumefantrine in healthy volunteers: a two-panel, two-way, two-period, randomized trial. HIV Med. 2013 Aug;14(7):421-9. doi: 10.1111/hiv.12019. Epub 2013 Feb 26. PMID 23441978